CLINICAL TRIAL: NCT05622734
Title: VOCALE LBD+ Leveraging Social Technologies and Problem-Solving Skills to Enhance Mastery Among Caregivers of Persons With Lewy Body Dementia
Brief Title: VOCALE LBD+ for Caregivers of Persons With Lewy Body Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Emory University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Oleg Zaslavsky, Associate Professor, School of Nursing, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00015485; P30AG064200 (NIH)
Record Dates: First submitted 2022-11-09; First posted 2022-11-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Caregiver Burden; Lewy Body Disease; Stress; Skill, Coping
MeSH Terms: conditions — Caregiver Burden; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOCALE LBD+ (Experimental)
  Interventions: Behavioral: VOCALE LBD+

INTERVENTIONS:
Behavioral: VOCALE LBD+ — Intervention employs a web-based platform that allows participants to engage asynchronously in an eight-week online intervention involving didactic training, peer-to-peer support, and moderated problem-solving skill enactment.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, acceptability, and initial efficacy of the VOCALE LBD+ intervention in caregivers of persons living with Lewy Body Dementia. The main question[s] it aims to answer are:

* What is the extent to which the VOCALE LBD+ intervention affects caregiving mastery scores at the end of the eight-week intervention
* What is the extent to which a change in caregiving mastery scores is retained four weeks after the end of the VOCALE LBD+ intervention

Participants will be asked to participate in a fully online asynchronous VOCALE LBD+ intervention that involves a moderated web-based discussion platform, peer-to-peer support, didactic training, and problem-solving skill enactment.

ELIGIBILITY:
Inclusion Criteria:

* Informal and/or lay caregiver of a patient with LBD
* Can read, write, and speak English
* Has access to a device that can be used for videoconferencing and/or phone calls
* 18 years or older

Exclusion Criteria:

* Not an informal and/or lay caregiver
* Cannot read and write in English
* No access to a device that can be used for videoconferencing and/or phone calls Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Zaslavsky, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VOCALE LBD+
Started | 39
Completed | 29
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | VOCALE LBD+
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 37
  More than one race | 1
  Unknown or Not Reported | 1
Spouse/partner [Count of Participants; unit: Participants] | 34

OUTCOME MEASURES:

1. Primary Outcome: Effect Size of Change From Baseline Caregiving Mastery at 4 Weeks
Description: Change in Pearlin's Caregiver Competence Scale Over Time, scale ranges from 7 to 35 with lower score indicating better mastery
Time Frame: Baseline; 4 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | VOCALE LBD+
Number analyzed (Participants) | 32
score on a scale | -0.04 [-0.36 to 0.29]

ADVERSE EVENTS:
Time Frame: Baseline to one month after the end of the intervention
Arm/Group | VOCALE LBD+
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05622734/Prot_SAP_000.pdf